CLINICAL TRIAL: NCT05627115
Title: Response Adapted Incorporation of Tislelizumab Into the Front-line Treatment of Older Patients With Hodgkin lYmphoma (RATiFY)
Brief Title: Response Adapted Incorporation of Tislelizumab Into the Front-line Treatment of Older Patients With Hodgkin lYmphoma
Acronym: RATiFY
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL 143242; 2022-003677-37 (EudraCT Number)
Record Dates: First submitted 2022-11-07; First posted 2022-11-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — tislelizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab Response-Adapted Treatment (Experimental): All patients will receive 3 cycles of tislelizumab 200 mg (IV) every 21 days. They will then undergo a PET-CT scan (PET1).
  Subsequent treatment with further tislelizumab, radiotherapy, and between 2-6 cycles of chemotherapy (Doxorubicin, Vinblastine, and Dacarbazine - AVD) is determined by the patient's stage and response at PET1.
  Interventions: Drug: Tislelizumab, AVD, Radiotherapy

INTERVENTIONS:
Drug: Tislelizumab, AVD, Radiotherapy — GROUP A: Early stage disease without adverse features in CMR: 2 further cycles tislelizumab then radiotherapy then 200mg IV tislelizumab once every 3 weeks until a maximum of 2 years total treatment. PET-CT (PET2) 12 weeks after radiotherapy.
  GROUP B: Early stage disease with adverse features in CMR: 2 cycles of AVD plus tislelizumab then radiotherapy. PET-CT (PET2) 12 weeks after the completion of radiotherapy.
  GROUP C: All early stage disease not in CMR: 4 cycles of AVD plus tislelizumab then PET-CT and radiotherapy. PET-CT 12 (PET2) weeks after radiotherapy.
  GROUP D: Advanced stage disease in CMR: 4 cycles of AVD plus tislelizumab then radiotherapy at investigator's discretion. PET-CT (PET2) 12 weeks after radiotherapy.
  GROUP E: Advanced stage disease not in CMR: 6 cycles of AVD plus tislelizumab then PET-CT then radiotherapy at investigator's discretion. PET-CT (PET2) 12 weeks after radiotherapy.
  Other Names: Response-adapted incorporation of tislelizumab

SUMMARY:
The goal of this clinical trial is to test the effect of tislelizumab treatment in patients with Hodgkin lymphoma. The main question it aims to answer is whether including a drug called tislelizumab in first-line treatment of Hodgkin lymphoma for patients age 60 years and older is effective and well-tolerated.

Participants will initially receive tislelizumab infusion every 21 days for 3 doses. After this a PET scan will be performed to assess the response. The subsequent treatment patients receive will depend on the following factors:

1. The lymphoma stage (early stage or advanced stage)
2. The presence or absence of specific high-risk features at the time of diagnosis
3. How well the lymphoma responds to the initial 3 doses of tislelizumab

DETAILED DESCRIPTION:
Trial patients who are deemed eligible for the trial will receive 3 cycles of tislelizumab which will be administered at a dose of 200 mg (IV) on day 1 of each 21-day cycle. Patients will then undergo a PET-CT scan (PET1). Subsequent treatment is determined by the patient's stage and response to tislelizumab (as determined by PET1).

Patients with early stage lymphoma and no high-risk features who respond very well to the initial 3 doses of tislelizumab will receive a further 2 doses of tislelizumab, followed by radiotherapy, followed by tislelizumab once every 21 days for up to 2 years.

All other patients will receive a combination of tislelizumab with chemotherapy for between 2 and 6 cycles. Each cycle will last 28 days. Tislelizumab will be given on day 1 and chemotherapy (doxorubicin (also known as Adriamycin), vinblastine and dacarbazine, or AVD) will be given on days 1 and 15, as injections or infusions into a vein. Following this some patients may require radiotherapy depending on their response to treatment.

Patients who are in complete metabolic response (CMR) at PET1 will receive 2 fewer cycles of tislelizumab and AVD therapy than those not in CMR.

A further 1 or 2 PET scans will be performed to assess how well the lymphoma has responded to the trial treatment, depending on the results of previous scans. After completing the treatment patients will then be followed-up for at least 2 years from the start of their participation in the trial.

Note: Initial patients will be recruited to a safety run in. Once 6 evaluable patients have completed 2 cycles of tislelizumab and AVD after PET1 the independent data monitoring committee (IDMC) will review the data, and if considered tolerable, recruitment will continue to the full sample size (80 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed untreated classic Hodgkin lymphoma (Stage I-IV)
2. Age 60 years or over
3. In the view of the investigator, fit for combination chemotherapy (includes those who would require planned dose reduction although no lower than 50% doxorubicin)
4. Written informed consent
5. Measurable disease on contrast enhanced CT as defined by Cheson et al., 2014 1 (Nodal lesion of longest diameter 1.5 cm or extranodal lesion of longest diameter 1.0 cm).
6. ECOG performance status 0-2
7. Adequate bone marrow function (Platelets ≥ 75 x 109/L without platelet transfusion for 72 hours, Neutrophils ≥ 1.0 x 109/L without G-CSF for 7 days)
8. Adequate liver function tests (ALT / AST ≤ 2.5 x ULN, total serum bilirubin ≤ 1.5 x ULN)
9. Creatinine Clearance ≥ 30 ml/min as defined by the Cockroft-Gault equation
10. Adequate cardiac function as determined by a transthoracic echocardiogram demonstrating left ventricular ejection fraction is ≥ 50% and confirming the absence of severe valvular heart disease
11. Willing to comply with the contraceptive requirements of the trial
12. Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

1. Nodular lymphocyte predominant Hodgkin lymphoma
2. History of autoimmune disorders (with the exception of hypothyroidism, type 1 diabetes, vitiligo, alopecia)
3. History of solid organ transplant
4. Grade 2 or higher peripheral neuropathy
5. Presentation with disease causing symptomatic compression of vital structures (e.g. stridor due to tracheal compression). Other cases of radiological compression of vital structures require discussion with TMG prior to registration
6. Women who are pregnant or breastfeeding
7. Active hepatitis B or C infection defined by

   1. Hepatitis B surface antigen positivity OR
   2. Anti-hepatitis B core antibody positivity with detectable circulating HBV DNA (hepatitis B core antibody patients with undetectable circulating HBV DNA are eligible but must take suitable prophylaxis for reactivation)
   3. Anti-Hepatitis C antibody positivity unless patient has been treated for hepatitis C and has undetectable HCV RNA
8. Known HIV infection
9. Positive PCR for SAR-CoV-2 RNA within the 2 weeks prior to registration. Patients with a history of SARS-CoV-2 are required to have a documented negative PCR swab since documented SARS-CoV-2 infection
10. Immunosuppressive therapy within the 2 months prior to registration apart from inhaled, intranasal or topical corticosteroids. Systemic corticosteroids are permitted prior to study entry but must be weaned to 10 mg prednisolone / day for a minimum of 7 days prior to cycle 1 day 1
11. Live vaccine given within 30 days prior to registration
12. Active infection requiring systemic therapy with ongoing symptoms at registration or where the planned duration of therapy would continue beyond cycle 1 day 1
13. Major surgery within 4 weeks prior to registration (excisional biopsy is not considered major surgery)
14. Myocardial infarction, unstable angina, coronary artery bypass graft, cerebrovascular accident or transient ischaemic attack within 6 months prior to registration
15. Previously treated haematological malignancy
16. Solid-organ malignancy active within the last 3 years, except where the natural history or treatment does not have the potential to interfere with assessment of safety or efficacy of trial treatment, for example:

    1. Adequately treated non-melanoma skin cancer considered to be in remission
    2. Melanoma in situ following resection
    3. Carcinoma in situ of the breast or cervix
    4. Carcinoma of the prostate of Gleason grade 6 or less with stable prostate-specific antigen levels
    5. Cancer considered cured by surgical resection or unlikely to impact survival in the next 3 years, for example local transitional carcinoma of the bladder or benign tumours of the adrenal gland or pancreas
17. A history of other malignancies should be discussed with the trial management group prior to registration
18. Patient not fit for AVD chemotherapy in the opinion of the investigator

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Two-year event-free survival (EFS) | 2 years after start of treatment
  To determine the effect of tislelizumab on 2 year EFS using a response-adapted approach to treatment in the front-line treatment of older patients with Hodgkin lymphoma

SECONDARY OUTCOMES:
The number / percentage of patients with the worst grade of each adverse event | From signing of informed consent until 30 calendar days post last IMP or post last investigational treatment administration (or after this date if the site investigator feels the event is related to an IMP and/or investigational treatment)
  To assess the safety and tolerability of tislelizumab alone and in combination with AVD. Worst grades will be calculated and presented as the number/percentage of patients with each event.
PET-defined response rates | After 3 cycles of tislelizumab (PET1) and at the end of the initial treatment (PET2) - up to 2 years after start of treatment
  To determine the effect of single agent tislelizumab on response (overall response rate (ORR), partial response (PR), complete response (CR) and Indeterminate Response (IR)) after 3 cycles of tislelizumab (PET1) and at end of initial treatment (PET2)
Overall survival (OS) of the whole population | From the date of registration until the date of death (any cause) or the date last seen (patients alive at time of analysis).
  To determine the effect of response adapted treatment with tislelizumab on OS
Progression free survival (PFS) of the whole population | 2 years after start of treatment
  To determine the effect of response adapted treatment with tislelizumab on PFS
EFS in early versus late stage patients | Up to 2 years after start of treatment
  To determine the effect of response adapted treatment with tislelizumab on EFS within early and late stage subgroups of patients
EFS in interim PET negative and positive patients | Up to 2 years after start of treatment
  To determine the effect of response adapted treatment with tislelizumab on EFS in PET1 negative and positive patients
Quality of life (QoL) assessed using EQ-5D-5L and FACT-Lym | From baseline until 2 years after start of treatment
  To assess the effect of treatment on QoL using using EQ-5D-5L and FACT-Lym at baseline and at multiple points during treatment and follow-up. These will be analysed using repeated measures including patient group.
Time to treatment failure | From the date of registration until the first date of progression, death or unplanned Hodgkin lymphoma therapy (switch to other regimens or any unplanned consolidation treatment) up to 2 years after start of trial treatment.
  To assess the rate of unplanned Hodgkin lymphoma therapy using Kaplan-Meier survival analysis, with plots and rates at 2 years presented.
PFS in early versus late stage patients | 2 years after start of treatment
  To determine the effect of response adapted treatment with tislelizumab on PFS within early and late stage subgroups of patients
OS in early versus late stage patients | Up to 2 years after start of treatment
  To determine the effect of response adapted treatment with tislelizumab on OS within early and late stage subgroups of patients
PFS in interim PET negative and positive patients | Up to 2 years after start of treatment
  To determine the effect of response adapted treatment with tislelizumab on PFS in PET1 negative and positive patients
OS in interim PET negative and positive patients | Up to 2 years after start of treatment
  To determine the effect of response adapted treatment with tislelizumab on OS in PET1 negative and positive patients
Frailty assessed using the Clinical Frailty Score (CFS) | From baseline until up to 2 years after start of treatment
  To assess the effect of treatment on frailty using the Clinical Frailty Score at baseline and at multiple points during treatment and follow-up. These will be analysed using repeated measures including patient group.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Graham Collins, Principal Investigator — Oxford University Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CR UK & UCL Cancer Trials Centre — http://www.ctc.ucl.ac.uk